CLINICAL TRIAL: NCT05524675
Title: The Effect of Multiple Medications on the Incidence of Organic Dyspepsia：a Prospective Observational Cohort
Brief Title: The Effect of Multiple Medications on the Incidence of Organic Dyspepsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, professor, Air Force Military Medical University, China
Other Study IDs: KY20222180-F-2
Record Dates: First submitted 2022-08-20; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dyspepsia is a very common gastrointestinal disease, presented as predominant symptom of upper abdominal pain. Underlying causes for dyspepsia can classified as organic or functional dyspepsia. Some medications (eg. non-steroid anti-inflammatory drugs (NSAIDs)) were associated with higher frequent incidences of organic lesions. Multiple medications showed an increased trend with aging of the population and multimorbidity. Multiple medications were suggested to be strongly relate to adverse drug events (ADEs), adverse drug reactions (ADRs), drug-drug interactions, and drug-disease interactions, which had been reported to lead to higher incidences of some diseases, including fractures, cognitive impairment and malnutrition. However, it was unknown if multiple medications was associated with more incidences of organic dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years old
2. patients who met broad criteria of dyspepsia
3. undergoing upper endoscopy and abdominal ultrasonography within one year.

Exclusion Criteria:

1. organ failure defined by Marshall standard
2. severe psychiatric illnesses
3. suspected or identified bowel obstruction
4. known malignancy
5. pregnancy or lactation
6. unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years old who met broad criteria of dyspepsia with upper endoscopy and abdominal ultrasonography within one year were eligible for our study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
the rate of patients diagnosed with organic upper gastrointestinal (GI) diseases. | 1 day
  All included patients underwent upper GI endoscopy and abdominal ultrasound and H. Pylori test. Barrett's esophagus, esophageal candidiasis, esophageal cancer, gastric ulcer, gastric erosion, gastric cancer, duodenal ulcer, duodenal erosion, cholecystitis, pancreatitis and biliary stones were classified as organic upper GI diseases.

SECONDARY OUTCOMES:
Functional dyspepsia | 6 months
  Functional dyspepsia was defined by Rome IV criteria, which was based on symptom and duration rather than scores. Patients diagnosed as Rome IV criteria met one or more of following criteria: postprandial fullness, early satiation, epigastric pain, and epigastric burning that are unexplained after a routine clinical evaluation, Criteria fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis. the above symptoms and durations were included in the questionaire. Physiological parameter was not required for Rome IV criteria.
Number of participants with different subtypes of functional dyspepsia | 6 months
  Functional dyspepsia was based on Rome IV criteria, which was based on symptom and duration rather than scores. Functional dyspepsia was classified into three subgroups：(1) Postprandial Distress Syndrome, Must include one or both of the following at least 3 days per week: 1. Bothersome postprandial fullness (ie, severe enough to impact on usual activities) 2. Bothersome early satiation (ie, severe enough to prevent finishing a regular-size meal) (2) Bothersome epigastric pain, Must include at least 1 of the following symptoms at least 1 day a week: 1. Bothersome epigastric pain (ie, severe enough to impact on usual activities) AND/OR 2. Bothersome epigastric burning (ie, severe enough to impact on usual activities). (3) mixed syndrome, defined when postprandial distress syndrome and epigastric pain syndrome presented simultaneously
Short Form of Nepean Dyspepsia Index (SF-NDI) | 1 day
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Hospital anxiety scale | 1 day
  Anxiety of patients are assessed by using Hospital Anxiety Scale.It contains 7 items, which assess symptoms experienced during the past week on a 0-3 scale. A subscore of > 8 for anxiety would indicate a clinical case.
Hospital depression scale | 1 day
  Depression of patients are assessed by using Hospital Depression Scale. It contains 7 items, which assess symptoms experienced during the past week on a 0-3 scale. A score of > 8 for depression would indicate a clinical case.
Quality of Life scores | 1 day
  Quality of Life scores assessed by Patient-reported outcomes measurement information system (PROMIS) Global-10 questionnaire.PROMIS Global-10 is a newly validated 10-question survey used to assess health care-related quality of life measures for the general population. It's a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient and a better quality of life.
Severity of functional dyspepsia judged by patients | 1 day
  Patients rated the severity of functional dyspepsia as mild, moderate, and severe by themselves.
Number of participants with other functional gastrointestinal diseases | 1 day
  Other functional gastrointestinal diseases#such as irritable bowel syndrome(IBS) or functional heartburn#etc.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xijing 986 Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi